CLINICAL TRIAL: NCT02839356
Title: Epinephrine Sprayed on the Papilla for the Prevention of Post-ERCP Pancreatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Epinephrine001
Record Dates: First submitted 2016-07-18; First posted 2016-07-21 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-07

CONDITIONS: Post-ERCP Acute Pancreatitis
MeSH Terms: interventions — Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug: epinephrine (Experimental): 20-mL irrigation with epinephrine diluted to 0.02% in saline over the entire papilla
  Interventions: Drug: epinephrine
- Drug: normal saline (Placebo Comparator): 20-mL irrigation with physiological saline over the entire papilla
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: epinephrine — 20-mL irrigation with epinephrine diluted to 0.02% in saline over the entire papilla
  Arms: Drug: epinephrine
Drug: normal saline — 20-mL irrigation with physiological saline over the entire papilla
  Arms: Drug: normal saline

SUMMARY:
Post-endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis (PEP) has been a well-recognized complication with significant morbidity and even mortality. A variety of possible mechanisms has been suggested in the occurrence of pancreatitis, but papillary edema caused by manipulations during cannulation or endoscopic treatment has received the most attention. The papillary edema may cause temporary outflow obstruction of pancreatic juice, and then increase ductal pressure, resulting in the occurrence of pancreatitis. Topical application of epinephrine on the papilla may reduce papillary edema. Moreover, it is reported that epinephrine sprayed on the papilla may be effective to prevent PEP. However, it is still unclear that epinephrine sprayed on the papilla can prevent acute pancreatitis after endoscopic retrograde cholangiopancreatography. We therefore designed a prospective randomized trial to determine whether epinephrine sprayed on the papilla prevent PEP after ERCP.

DETAILED DESCRIPTION:
Between July 2016 and December 2017, 670 consecutive patients older than 18 years who are scheduled to undergo diagnostic or therapeutic ERCP at the Anhui Provincial Hospital will be recruited for the study. Patients were randomized using opaque, sealed envelopes containing random numbers assigning them to undergo a spray of epinephrine (epinephrine group) or saline (control group) on the major papilla. A two proportion equality test will be conducted to explore whether incidence rates are different. Descriptive statistics including number (N), mean, median, standard deviation, minimum and maximum, will be produced for all continuous variables. Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age > 18 years.
2. Normal amylase level before undergoing ERCP.
3. Signed inform consent form and agreed to follow-up on time.

Exclusion Criteria:

1. Pregnancy or history of allergy to epinephrine.
2. Medical or psychological condition that would not permit the patient to complete the study or sign the informed consent.
3. Patients involved in other study within 60 days.
4. Billroth II or Roux-en-Y anatomy
5. Acute pancreatitis.
6. All contraindications to epinephrine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The prophylaxis effect of epinephrine sprayed on the papilla on post-ERCP pancreatitis | PEP occurence rate at 24 h after ERCP in two groups.
  If the serum amylase of patients elevation and 3 times higher than the normal values after ERCP 24 hours in high risk patients, who also have clinical symptoms, without other acute abdominal diseases,such as gastrointestinal perforation,acute cholecystitia and acute cholangitis and etc. In this condition, it will be defined PEP(post-ERCP pancreatitis). Descriptive statistics will be produced for all continuous variables. Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.
  Descriptive statistics will be produced for all continuous variables. Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.

SECONDARY OUTCOMES:
Compare epinephrine group with control group on the incidence of hyperamylasemia/adverse events. | the incidence of hyperamylasemia/adverse events at 24 h after ERCP in two groups
  Hyperamylasemia will be defined as the serum amylase 3 times more than the upper normal values, without clinical symptoms. During the study, any unexpected medical issue will be called adverse event.
  Descriptive statistics will be produced for all continuous variables. Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Shao Feng, MD, Study Director — Department of General Surgery, Anhui Provincial Hospital Affiliated with Anhui Medical University
Locations (1):
- Department of General Surgery, Anhui Provincial Hospital Affiliated with Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No